CLINICAL TRIAL: NCT02035800
Title: Bone Resorption, Osteoclastogenesis and Adalimumab
Acronym: BROCAII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMM 11-0163
Record Dates: First submitted 2013-12-10; First posted 2014-01-14 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid Arthritis; Adalimumab; Humira
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adalimumab (humira) (Experimental): As standard of care.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Patient will received medication as standard of care
  Other Names: Humira

SUMMARY:
Broca II is the prolongation of the original study name BROCA. In BROCA study, only 25 patients participated and it was not enough to concluded clearly our hypothesis.

DETAILED DESCRIPTION:
Osteoclasts (OC) are clearly involved in joint destruction in Rheumatoid Arthritis (RA), as shown by clinical and experimental data. Tumor Necrosis Factor Alpha (TNF-alpha), a major pathologic mediator in RA, may induce bone resorption either directly, stimulating osteoclastogenesis or indirectly, by influencing receptor activator of nuclear factor kappa-B ligand (RANKL), osteoprotegerin (OPG) and prostaglandin production by osteoblasts. Anti-TNF agents reduce bone destruction in RA but their effects on osteoclast biology in patients with RA are little known.

The original BROCA study, which included a cohort of 25 RA patients, aimed to study the effect of treatment with Adalimumab on times zero, 3 and 6 months on the following osteoclastic parameters: 1) the number of osteoclast precursor (CD14+) cells in the peripheral blood, 2) the number of osteoclasts generated in vitro, and 3) the amount of bone resorption in vitro before, 3 and 6 months after treatment with Adalimumab. The secondary outcomes were 1) The effect of treatment with Adalimumab on disease activity score defined as a DAS28 score (Disease Activity Score, 2) The effect of treatment with Adalimumab (also name: Humira) on change in functional status by the health assessment questionnaire (HAQ), and 3) Parallel in vitro differentiation assays (number of osteoclasts generated and amount of bone resorption) in the presence of exogenous Adalimumab in the concentration range found in the plasma of treated patients to detect a direct effect of the medication in vitro in osteoclastogenesis.

The results showed that treatment with Adalimumab induced a statistically significant reduction in the clinical scores DAS28 and HAQ, as has been shown by many clinical studies . Even though no statistically significant effect of the treatment was found on the number of osteoclast precursors, the number of osteoclasts generated in vitro or the surface of bone resorption in vitro, there was a clear trend towards a decrease in the last two parameters. We believe this lack of statistical significance is due to a type II error, a consequence of the much higher variance of the primary parameter (number of in vitro-generated osteoclasts) in the patient cohort than we could foresee from the initial data from normal donors. Moreover, there was a statistically significant correlation (p=0.416, linear regression) between the difference in the number of osteoclasts in time zero and six months and the difference in the HAQ score, which not only supports the hypothesis that the treatment with Adalimumab may be associated with a reduction in the number of osteoclasts but also suggests that this reduction may be associated with a better response to the treatment. The general objective of the proposed prolongation of the BROCA study is to verify these two working hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 18 and over,
* Satisfying the 1987 American College of Rheumatology (ACR) criteria for RA
* Receiving a prescription of Adalimumab 40 mg subcutaneous every two weeks.

Exclusion Criteria:

* Patients not capable or willing to provide informed consent
* Patients starting Adalimumab less than five half-lives after the interruption of a previous anti-TNF therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Verify if the treatment with Adalimumab may be associated with a reduction in the number of osteoclasts. | 6 months after treatment
  By calculating the number of osteoclast and osteoblast in patient serum.

SECONDARY OUTCOMES:
Verify if this reduction may be associated with a better response to the treatment. | 6 months after treatment
  Disease activity defined as a DAS28 score
To verify reduction of osteoclasts may be associated with a better response to the treatment. | 6 months after treatment
  Functional status by the HAQ
To verify reduction of osteoclasts may be associated with a better response to the treatment. | 6 months after traitment
  Radiological progression defined by Sharp scores

CONTACTS AND LOCATIONS:
Overall Officials: Artur Ferandnes, Principal Investigator — Centre de recherche Étienne Le-Bel at Centre hospitalier universitaire de Sherbrooke
Locations (1):
- CRC Étienne Le-Bel at CHUS, Sherbrooke, Quebec, Canada